CLINICAL TRIAL: NCT04455984
Title: Multimodality Treatment Including Curative Resection of Advanced Stage Non-small Cell Lung Cancer - an Explorative, Retrospective Pilot Study
Brief Title: Multimodality Treatment Including Curative Resection of Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katharina Sinn, MD, Medical University of Vienna
Other Study IDs: 193132122
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Advanced Non-small-cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemoradiotherapy: Patients with advanced NSCLC treated with neoadjuvant platinum-based chemoradiotherapy followed by curative-intent surgery
  Interventions: Other: Date collection
- Neoadjuvant chemotherapy: Patients with advanced NSCLC treated with neoadjuvant platinum-based chemotherapy followed by curative-intent surgery
  Interventions: Other: Date collection

INTERVENTIONS:
Other: Date collection — Retrospective data analysis

SUMMARY:
This study retrospectively evaluates clinical parameters and outcome of patients with advanced stage non-small cell lung cancer treated with neoadjuvant therapy followed by curative-intent surgery at the Divison of Thoracic Surgery at the Medical University of Vienna

DETAILED DESCRIPTION:
This study will be undertaken as a retrospective cohort study at Devision of Thoracic Surgery, Medical University of Vienna. All patients with non-small-cell lung cancer, who received an induction chemo- or chemoradiotherapy followed by surgery in a curative intention at the Devision of Thoracic Surgery, Medical University, will be included. The aim of this study is to evaluate peri- and postoperative clinical parameters and short- and long-term outcomes in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced NSCLC and multimodality treatment including curative-intent resection

Exclusion Criteria:

* Patients with early stage NSCLC
* Patients with advanced NSCLC without multimodality treatment
* Patients without curative resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with non-small-cell lung cancer, who received an induction chemo- or chemoradiotherapy followed by surgery in a curative intention at the Devision of Thoracic Surgery, Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 18 years
  * Overall survival of stage III NSCLC in resectable patients undergoing induction treatment and curative intent surgery
  * Overall survival of stage III NSCLC in resectable patients undergoing induction treatment and curative intent surgery
  * Overall survival of stage III NSCLC in resectable patients undergoing induction treatment and curative intent surgery Overall survival of stage III NSCLC in resectable patients undergoing induction treatment and curative intent surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No